CLINICAL TRIAL: NCT02110264
Title: Depot Pharmacotherapies for Opioid-Dependent Offenders: Outcomes and Costs
Brief Title: Injectable Pharmacotherapy for Opioid Use Disorders (IPOD)
Acronym: IPOD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA034743
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Opioid Use Disorders
Keywords: Opioid Use; Incarceration; Vivitrol; Patient Navigator; Drug Education
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vivitrol (XR-NTX) (Experimental): 50 participants will be randomized to the long-acting naltrexone condition (XR-NTX) which will include monthly injections of study drug.
  Interventions: Drug: XR-NTX
- XR-NTX+PN (Experimental): 50 participants will be randomized to receive long-acting naltrexone (XR-NTX) and will be assigned to a patient navigator (PN).
  Interventions: Drug: XR-NTX; Behavioral: XR-NTX+PN
- ETAU (Active Comparator): 50 participants will be randomized to the drug-education/treatment-as-usual group.
  Interventions: Behavioral: ETAU

INTERVENTIONS:
Drug: XR-NTX — Monthly injections of XR-NTX will be administered to participants assigned to either the XR-NTX or XR-NTX+PN groups.
  Other Names: long-acting naltrexone; Vivitrol
  Arms: Vivitrol (XR-NTX); XR-NTX+PN
Behavioral: XR-NTX+PN — In addition to long-acting naltrexone (XR-NTX), participants assigned to the XR-NTX+PN condition will meet regularly with a patient navigator to assist in accessing psychosocial services when released from jail.
  Other Names: Patient Navigator
  Arms: XR-NTX+PN
Behavioral: ETAU — Participants assigned to the ETAU group will receive drug education.
  Other Names: Treatment-as-usual; Drug Education
  Arms: ETAU

SUMMARY:
The aim of this trial is to assess the clinical utility, effectiveness, and cost implications of treatment for incarcerated offenders with opioid use disorders who are randomly assigned to one of three treatment conditions to include a depot formulation of naltrexone (XR-NTX, as Vivitrol®) only (XR-NTX), Vivitrol provided with sessions with a patient navigator (PN) XR-NTX+PN, and a drug education procedure (ETAU) before being released to the community. This trial will investigate whether effective medication therapy used in non-incarcerated populations will also be effective in incarcerated individuals. Empirical evidence demonstrates that starting treatment before release greatly increases the probability of successful outcome including reduced alcohol and drug use, increased employment rates, and reduced recidivism rates.

DETAILED DESCRIPTION:
This randomized, open-label trial will examine the feasibility, efficacy, and net economic benefits of XR-NTX for opioid addiction delivered with and without a platform of PN provided for six months compared against an education (ETAU) condition. Before release from jail, participants in the XR_NTX and XR-NTX+PN conditions will receive their first Vivitrol injection (and those in the XR-NTX+PN condition will meet with a Patient Navigator) and will then be scheduled for medication management sessions twice monthly for months 1-3, with monthly injections in months 4-6. Participants in the XR-NTX+PN condition will meet with a PN who will provide behavioral assistance to overcome possible barriers to community outpatient treatment and will be provided with referrals for community treatment programs. Participants in the ETAU condition will receive education designed to reduce the likelihood of overdose on the same schedule as the XR-NTX and XR-NTX+PN groups.

Participants will be individuals who meet DSM-5 (Diagnostic and Statistical Manual-5) (via CIDI-2 (composite international diagnostic interview

)) criteria for opioid use disorders, are 18 years and older, who have been detoxified from opioids in the Metropolitan Detention Center in Albuquerque, New Mexico. This study will include only those participants for whom the study physician determines that possible treatment with the study drug is in the best interest, and informed consent will be obtained.

All participants will be scheduled for twice-monthly medical management and assessment appointments for the first three months of the 24-week post-release intervention phase, with monthly appointments for months 4-6. Eligible participants will be randomly assigned to treatment condition (XR-NTX, XR-NTX+PN, ETAU) in equal numbers. XR-NTX and XR-NTX+PN participants will undergo a naloxone challenge to ensure opioid abstinence at the time of Vivitrol induction. Those in the XR-NTX+PN condition will be provided with a PN (patient navigator) who will facilitate attendance at outpatient treatment programs as well as assist with other needs. The ETAU group will not receive any medication but will be scheduled for assessments and education on drugs of abuse, maintaining abstinence, and methods for avoiding overdoses on the same schedule as the other two groups. All groups will also be provided with referrals to community-based substance abuse treatment programs.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age or older,
2. Meet criteria for DSM-5 opioid use disorders,
3. Be detained for at least 48 hours,
4. Have an expected release date within one year,
5. Plan to reside in area after release.

Exclusion Criteria:

1. Have a medical (e.g., liver failure, congestive heart failure) or psychiatric condition (e.g., suicidal ideation, psychosis) that would make participation unsafe in the judgment of the medical staff or the PI,
2. Have current or chronic pain or have plans to undergo pain treatment/therapy,
3. Have known sensitivity to naltrexone or naloxone,
4. Have participated in an investigational drug study within the past 30 days prior to screening,
5. Be a nursing or pregnant female, or not agree to use a medically acceptable form of birth control such as oral contraceptives, barrier (diaphragm or condom), levonorgestrel implant, intra-uterine progesterone contraceptives system, medroxyprogesterone acetate contraceptive injection, or complete abstinence. Females who become pregnant during the course of the study will be withdrawn from the study and, if requested, will be provided with referrals for drug treatment and/or medical care,
6. Have any pending legal action that could prohibit continued participation for the 24-week intervention period of the study, such as legal proceedings that could possibly result in incarceration,
7. Have a current pattern of alcohol, benzodiazepine, or other depressant or sedative hypnotic use, as determined by the study physician which would preclude safe participation in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Farabee, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of New Mexico Center on Alcoholism, Substance Abuse and Addictions, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Farabee D, Hillhouse M, Condon T, McCrady B, McCollister K, Ling W. Injectable pharmacotherapy for opioid use disorders (IPOD). Contemp Clin Trials. 2016 Jul;49:70-7. doi: 10.1016/j.cct.2016.06.003. Epub 2016 Jun 6. PMID 27282118

RESULTS

PARTICIPANT FLOW:
Groups:
- Vivitrol (XR-NTX): Long-acting naltrexone condition (XR-NTX) which will included monthly injections of study drug.
- XR-NTX+PN: Long-acting naltrexone (XR-NTX) and assignment of a patient navigator (PN).
- ETAU: Treatment as usual, along with will receive drug education.
Period: Overall Study
Arm/Group | Vivitrol (XR-NTX) | XR-NTX+PN | ETAU
Started | 53 | 50 | 48
Completed | 35 | 38 | 39
Not Completed | 18 | 12 | 9

BASELINE CHARACTERISTICS:
Population: 16 participants were deemed ineligible because they were directly transferred from jail to prison.
Groups:
- Vivitrol (XR-NTX): Long-acting naltrexone condition (XR-NTX) which will include monthly injections of study drug.
- XR-NTX+PN: Long-acting naltrexone (XR-NTX) and assigned to a patient navigator (PN).
- ETAU: Drug-education/treatment-as-usual.
- Total: Total of all reporting groups
Arm/Group | Vivitrol (XR-NTX) | XR-NTX+PN | ETAU | Total
Number analyzed (Participants) | 46 | 45 | 44 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (9.5) | 34 (8.8) | 33 (9.7) | 33 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 14 | 37
  Male | 35 | 33 | 30 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 4 | 13
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 6 | 12
  White | 36 | 32 | 26 | 94
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 46 | 45 | 44 | 135

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use
Description: The primary objective is to compare outcomes of the three intervention groups, based on self-reports at 6-months post-intervention.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Vivitrol (XR-NTX): Long-acting naltrexone condition (XR-NTX) which included monthly injections of study drug.
Arm/Group | Vivitrol (XR-NTX) | XR-NTX+PN | ETAU
Number analyzed (Participants) | 37 | 42 | 41
Participants | 6 | 12 | 7

2. Secondary Outcome: Opioid Use Disorder
Description: Number of participants meeting DSM-5 OUD (opioid use disorder) criteria via modified CIDI-2 Substance Abuse Module
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol (XR-NTX) | XR-NTX+PN | ETAU
Number analyzed (Participants) | 37 | 42 | 41
Participants | 4 | 4 | 3

ADVERSE EVENTS:
Time Frame: 6 months for participants in either of the two medication conditions.
Description: AEs were systematically collected from participants in the two medication conditions.
Arm/Group | Vivitrol (XR-NTX) | XR-NTX+PN | ETAU
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/50 | 0/48
Other Adverse Events (participants affected / at risk) | 4/53 | 5/50 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vivitrol (XR-NTX) (N=53) | XR-NTX+PN (N=50) | ETAU (N=48)
Helpatobiliary disorder (Hepatobiliary disorders) | 0 | 1 | 0 — Abdominal pain, jaundice, abnormal liver enzymes
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vivitrol (XR-NTX) (N=53) | XR-NTX+PN (N=50) | ETAU (N=48)
Pain at injection site (General disorders) | 2 | 4 | 0
Precipitated withdrawal (Injury, poisoning and procedural complications) | 1 | 1 | 0
photophobia (Eye disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02110264/Prot_SAP_000.pdf